CLINICAL TRIAL: NCT00536094
Title: School-Based CBT for Anxious African-American Children
Brief Title: School-based Treatment for Anxious Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Golda S. Ginsburg, Ph.D., Professor, National Institute of Mental Health (NIMH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R34MH074552 (NIH); R34MH074552 (NIH); DSIR 84-CTS
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2012-04

CONDITIONS: Anxiety Disorders
Keywords: Cognitive behavioral therapy; Youth; School; African American
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive cognitive behavioral therapy for anxiety that includes exposure
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)
- 2 (Active Comparator): Participants will receive treatment as usual as delivered by school-based clinicians
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) — CBT includes 45-minute psychotherapy sessions once a week for a period of approximately 12 weeks.
  Other Names: CBT
  Arms: 1
Behavioral: Treatment as usual (TAU) — TAU includes 45-minute psychosocial treatment sessions once a week for a period of approximately 12 weeks.
  Other Names: TAU
  Arms: 2

SUMMARY:
This study will determine the effectiveness of a school-based cognitive behavior therapy in urban, predominantly low-income, African-American children diagnosed with an anxiety disorder.

DETAILED DESCRIPTION:
Anxiety disorders are among the most common childhood disorders. Although anxiety is a normal part of life and growing up, for some children this anxiety becomes chronic, relentless, and progressively worse if left untreated. Physical symptoms typically accompany the intense anxiety caused by the disorder and may include blushing, profuse sweating, trembling, nausea, and difficulty talking. Anxiety disorders among children have become increasingly prevalent, indicating that excessive fear, worry, and anxiety in children are emerging public health issues. Recent studies have shown that CBT is an effective form of treatment for childhood anxiety disorders; however, it often requires the use of expert CBT clinicians. The purpose of this study is to deliver a school-based version of CBT to predominantly low-income, inner-city, African-American children with anxiety disorders. Clinicians within the school will undergo CBT training and adapt the treatment program to fit the needs of the participating children.

All participants in this study will undergo an initial evaluation to assess anxiety symptoms, disorders, and associated impairments. The children will then be randomly assigned to receive 12 weekly sessions of school-based CBT or treatment as usual, which will involve 12 weekly sessions of psychosocial treatment. Three parent sessions will be offered for families in both groups at Weeks 2, 6, and 10. All treatment sessions will occur at school during the day and will be led by school-based clinicians. A follow-up session will be conducted at post-treatment and 1 month after the last session to assess anxiety symptoms and disorders. Parent, teacher, and clinician ratings will also be used to assess the treatment outcomes of each child.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for primary diagnosis of generalized anxiety disorder (GAD), social anxiety disorder (SAD), specific phobia (SP), or social phobia (SOP)
* Received a score of at least 4 on the ADIS for DSM-IV:C's Clinician's Severity Rating Scale (CSR) for GAD, SAD, SP, and/or SOP
* Received a minimum 1 point difference in ADIS for DSM-IV:C severity scores between the primary disorder and other disorders (e.g., depressive disorders, disruptive behavior disorders, attention deficit hyperactive disorder [ADHD], and other anxiety disorders such as obsessive compulsive disorder [OCD], post-traumatic stress disorder [PTSD], acute stress disorder)

Exclusion Criteria:

* Diagnosed with a pervasive developmental disorder, mental retardation, organic mental disorders, schizophrenia, or other psychotic disorders
* Psychotic or suicidal
* Currently receiving treatment for anxiety
* Requires immediate or alternative treatment
* Previously failed a trial of at least 10 sessions for anxiety within 2 years of study entry
* Absent 50% of school days in the 2 months preceding random assignment to treatment groups
* History of child abuse and requires ongoing Department of Social Services supervision

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2006-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule for DSM-IV: Child Version | Measured at pre-treatment, post-treatment, and one month follow-up

SECONDARY OUTCOMES:
Screen for Child Anxiety Related Disorders (SCARED) - Child Version | Measured at pre-treatment, post-treatment, and one month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Golda Ginsburg, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- [Background] Ginsburg, G. S., Becker, K. D., Kingery, J.,and Nichols, T. (2008). Transporting CBT for childhood anxiety disorders into inner city school-based mental health clinics. Cognitive and Behavioral Practice, 15, 148-158.